CLINICAL TRIAL: NCT04691206
Title: A Resident-initiated, Step-wise, Competency-based, Graduated Operative Curriculum to Enhance Resident Autonomy for Laparoscopic Cholecystectomy
Brief Title: Operative Curriculum Gallbladder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sarah A. McLaughlin, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-002606
Record Dates: First submitted 2020-10-17; First posted 2020-12-31 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Surgical Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- standardized step-wise operative curriculum (Other): General surgery residents at Mayo Clinic will complete surveys measuring resident autonomy, performance, confidence and case complexity at baseline and postoperatively following laparoscopic cholecystectomy to serve as a pre-intervention baseline.
  A standardized step-wise operative curriculum will then be implemented Residents will follow and graduate through this curriculum by initiating a perioperative model of briefing objectives, intraoperative teaching, and debriefing feedback (BID). The effectiveness of the intervention will then be measured by comparing survey results pre and post intervention.
  Interventions: Other: briefing objectives, intraoperative teaching, and debriefing feedback

INTERVENTIONS:
Other: briefing objectives, intraoperative teaching, and debriefing feedback — A standardized step-wise operative curriculum amongst general surgeons will be implemented among all general surgery residents. Residents will follow and graduate through this curriculum by initiating a perioperative model of briefing objectives, intraoperative teaching, and debriefing feedback (BID).

SUMMARY:
The goal of this study is to implement and evaluate the need, feasibility and effectiveness of a resident-initiated, step-wise, graduated operative curriculum designed to enhance resident autonomy for laparoscopic cholecystectomy for general surgery residents.

DETAILED DESCRIPTION:
The goal of this study is to improve resident autonomy and confidence through detailed and stepwise feedback and to also assess resident and attending perceptions regarding resident skill and autonomy.

ELIGIBILITY:
Inclusion Criteria:

* All Mayo Clinic general surgery residents and attendings across all campuses

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Surgical Resident's Autonomy | Baseline, postoperatively approximately one day
  Measured using a validated Zwisch based survey to compare the rate of progression of surgical resident autonomy performing laparoscopic cholecystectomy pre and post implementation of standardized step-wise operative curriculum
Change is Surgical Resident's Operative Skills | Baseline, postoperatively approximately one day
  Measured using a validated Zwisch based survey to compare the rate of progression of surgical resident operative skills performing laparoscopic cholecystectomy pre and post implementation of standardized step-wise operative curriculum
Change in Surgical Resident's Confidence | Baseline, postoperatively approximately one day
  Measured using a validated Zwisch based survey to compare the rate of progression of surgical resident reported confidence performing laparoscopic cholecystectomy pre and post implementation of standardized step-wise operative curriculum

SECONDARY OUTCOMES:
Difference in Surgical Resident and Attending Physician Perceptions | Baseline, postoperatively approximately one day
  Difference between surgical resident and attending physician's perceptions of progression of resident operative skills performing laparoscopic cholecystectomy pre and post implementation of standardized step-wise operative curriculum using a validated Zwisch based survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah McLaughlin, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials